CLINICAL TRIAL: NCT06952426
Title: A Mobile App-Based, Prospective, Observational Study to Evaluate Disease Burden and Treatment Patterns in Immunoglobulin A Nephropathy (IgAN) in the US
Brief Title: A Mobile App-Based Study to Evaluate Disease Burden and Treatment Patterns in Immunoglobulin A Nephropathy (IgAN) in the US
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023AUS02
Record Dates: First submitted 2025-02-26; First posted 2025-04-30 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Immunoglobulin A Nephropathy
Keywords: IgAN; HRQoL; Iptacopan; atrasentan; Immunoglobulin A nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — iptacopan; Atrasentan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Immunoglobulin A nephropathy (IgAN)-Iptacopan: IgAN patients taking iptacopan and their caregivers
  Interventions: Other: Iptacopan
- IgAN-atrasentan: IgAN patients taking atrasentan and their caregivers
  Interventions: Other: Atrasentan
- IgAN-other treatment: IgAN patients taking other specific treatment and their caregivers
  Interventions: Other: Other treatment
- IgAN-no treatment: IgAN patients taking none treatment and their caregivers
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Participants and their caregivers will report home reported outcomes (HRO) data on symptom burden to understand symptom variability and health-related quality of life (HRQoL).
  Groups: IgAN-no treatment
Other: Other treatment — Participants and their caregivers will report HRO data on symptom burden and treatment usage to understand symptom variability and HRQoL.
  Groups: IgAN-other treatment
Other: Iptacopan — Participants and their caregivers will report HRO data on symptom burden and treatment usage to understand symptom variability and HRQoL including those taking iptacopan.
  Groups: Immunoglobulin A nephropathy (IgAN)-Iptacopan
Other: Atrasentan — Participants and their caregivers will report HRO data on symptom burden and treatment usage to understand symptom variability and HRQoL including those taking atrasentan.
  Groups: IgAN-atrasentan

SUMMARY:
The study aims to longitudinally capture the full spectrum of symptoms, treatment utilization, and overall health-related quality of life (HRQoL) experienced by Immunoglobulin A nephropathy (IgAN) patients and their caregivers.

DETAILED DESCRIPTION:
This will be a prospective, observational study. Data will be collected using the Folia Health platform. Participation in the study will occur through use of the Folia mobile platform, where study participants will be directed to a study-specific platform environment to review and sign the consent form and enroll. Each participant will complete an initial 6-month study data collection period which includes home reported outcomes (HRO) tracking along with study specific components including a baseline survey, monthly check-in prompts, and endline study evaluation survey. After the 6-month period, participants can continue to use Folia to track their HROs for their own personal use. With their consent, the data they enter after the initial 6-month period may be reviewed for ongoing data integrations with Novartis APPRISE data platform for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IgAN, regardless of symptom or treatment history
* Adult aged 18 or older; adult caregiver to an adult patient aged 18 or older; or adult caregiver to a pediatric patient under 18 years of age
* US-based with a proficient understanding of and ability to read the English language

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve patients who has received Immunoglobulin A nephropathy diagnosis in US.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with IgAN specific symptoms | monthly up to month 6
  To assess and gain a comprehensive understanding of the patient-reported burden of Immunoglobulin A nephropathy (IgAN) using home-reported outcome (HRO) symptom tracking data. Patients will select from a list of suggested symptoms. The 10 symptoms most frequently reported will be presented and analyzed.
Average self-reported severity of each of these top 10 symptoms | monthly up to month 6
  To assess and gain a comprehensive understanding of the patient-reported burden of IgAN using HRO symptom tracking data.
Variability in self-reported severity of each of these top 10 symptoms | monthly up to month 6
  To assess and gain a comprehensive understanding of the patient-reported burden of IgAN using HRO symptom tracking data.

SECONDARY OUTCOMES:
Average temporal frequency of treatment administration, for each IgAN-specific treatment | monthly up to month 6
  To characterize IgAN treatment utilization patterns.
Number of participants by reason for skipping treatment | monthly up to month 6
  To identify participant reported reasons for skipping treatment.
Differences in symptom occurrence for participants in each treatment group | monthly up to month 6
  Symptom occurrence (number of participants who report it) between patients in each treatment group will be presented.
Differences in symptom severity for participants in each treatment group | monthly up to month 6
  Symptom severity between patients in each treatment group will be presented. Severity is measured on a 1-5 severity scale with higher numbers indicating more severe symptoms.
Differences in symptom frequency for participants in each treatment group | monthly up to month 6
  To compare symptom frequency (instances of a symptom's occurrences divided by the total number of tracks) patients in each treatment group will be presented.
Change in average symptom occurrence from pre-treatment to post-treatment utilization, for participants who initiated iptacopan or atrasentan during the study period | monthly up to month 6
  Change in symptom occurrence from pre- to post-iptacopan and/or atrasentan utilization, among patients receiving iptacopan and/or atrasentan.
Change in average symptom severity from pre-treatment to post-treatment utilization, for participants who initiated iptacopan or atrasentan during the study period | monthly up to month 6
  Change in symptom severity from pre- to post-iptacopan and/or atrasentan utilization, among patients receiving iptacopan and/or atrasentan.
Change in average symptom frequency from pre-treatment to post-treatment utilization, for participants who initiated iptacopan or atrasentan during the study period | monthly up to month 6
  Change in symptom frequency from pre- to post-iptacopan and/or atrasentan utilization, among patients receiving iptacopan and/or atrasentan.
Number of participants in each treatment group who are classified as having a high vs moderate vs low flare burden | monthly up to month 6
  To compare proportion of patients classified as high, moderate, or low flare burden between patients in each treatment group.
Change over time in monthly check-in responses assessing health-related quality of life (HRQoL), for participants in each treatment group | monthly up to month 6
  To compare change in monthly HRQoL between patients in each treatment group. HRQoL will be assessed qualitatively through survey questions at monthly timepoints (no PRO scale), and participants will report on missed work or school, satisfaction with treatment plan, and frequency and characteristics of patient-defined difficult days.
Patient-reported outcome (PRO) scores for participants in each treatment group - FACIT-F | monthly up to month 6
  To compare change in monthly PRO scores between patients in each treatment group. The Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F) is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. FACIT ranges from 0 to 52, with 0 being the worst possible score and 52 the best.
Patient-reported outcome (PRO) scores for participants in each treatment group - EQ-5D-5L | monthly up to month 6
  To compare change in monthly PRO scores between patients in each treatment group.
  The EQ-5D-5L consists of 2 items - a descriptive system and a visual analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS records the respondent's self-rated health on a 20-cm vertical, visual analogue scale numbered 0 to 100 with 100 meaning the best possible health.

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigational site, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No